CLINICAL TRIAL: NCT04601493
Title: PRescribing INterventions for Chronic Pain Via the Electronic Health Record Study - Opioid-Naive Population
Acronym: PRINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00006522-2; R33DA046084 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder; Opioid Use; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 43 Primary Care Clinics will be randomized to be in one of 4 arms: 1) Care as usual, 2) Choice architecture nudge, 3) Prescription Drug Monitoring Program (PMP) Integration & nudge, 4) Choice architecture nudge + PMP Integration & nudge
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Care as Usual (No Intervention): Clinics assigned to this arm will continue to care for the patients as usual in regards to opioid prescribing.
- Choice Architecture Nudge (Experimental): Clinics in this arm will receive the choice architecture nudge intervention.
  Interventions: Behavioral: Choice Architecture Nudge
- PMP Integration & Nudge (Experimental): Clinics in this arm will receive the Prescription Drug Monitoring (PMP) Integration & Nudge intervention.
  Interventions: Behavioral: PMP Integration & Nudge
- Choice Architecture Nudge + PMP Integration & Nudge (Experimental): Clinics in this arm will receive both the choice architecture nudge and prescription drug monitoring (PMP) integration & nudge interventions.
  Interventions: Behavioral: Choice Architecture Nudge; Behavioral: PMP Integration & Nudge

INTERVENTIONS:
Behavioral: Choice Architecture Nudge — During the choice architecture nudge intervention, Primary Care Providers (PCPs) will be sent alerts in the Electronic Health Record (EHR) system when they initiate an opioid order for a patient who has not had an opioid prescription within the past six months. The alert provides guidance language about opioid prescribing and prompts the PCP to open the "SmartSet" to order non-opioid treatment alternatives. PCPs can choose to ignore this, but opening the SmartSet is the default option. When the SmartSet is opened, PCPs can choose to click on a variety of treatment order options, including both non-opioid pharmacological options and non-pharmacological options (e.g., referral to physical therapy or pain clinic).
  Arms: Choice Architecture Nudge; Choice Architecture Nudge + PMP Integration & Nudge
Behavioral: PMP Integration & Nudge — During the Prescription Drug Monitoring Program (PMP) integration & nudge intervention, Primary Care Providers (PCPs) will have integrated access to the PMP embedded within the EHR. All clinicians can already access the PMP to look up a patient's prior opioid prescriptions and prescription fills. However, this process involves signing in to the separate PMP website and can be complicated and time-consuming within typical clinical workflow. The integrated PMP tool makes it much easier and faster for a PCP to access the PMP information for a given patient.
  Arms: Choice Architecture Nudge + PMP Integration & Nudge; PMP Integration & Nudge

SUMMARY:
The objective of this research is to assess the effects of electronic health record (EHR)-based decision support tools on primary care provider (PCP) decision-making around pain treatment and opioid prescribing. The decision support tools are informed by principles of "behavioral economics," whereby clinicians are "nudged," though never forced, towards guideline-concordant care.

DETAILED DESCRIPTION:
To test the effects of these decision support tools for improving the quality of care for pain treatment, the investigators will implement a pragmatic clinic-randomized trial across the primary care clinics of Fairview Medical Group and University of Minnesota Physicians.

The study has two parallel components. The decision support tools to be tested will differ somewhat depending on whether a given patient is opioid-naïve, or whether a given patient is a current opioid-user. Four sets of analyses will be conducted separately: one for the opioid-naïve group using EHR data, one for the current opioid-user group using EHR data, one at the PCP-level using web survey data, and one at the PCP-level using MN Prescription Drug Monitoring Program (PDMP) data.

ELIGIBILITY:
Inclusion Criteria:

- All primary care providers from all of the Fairview and University of Minnesota Physicians study clinics

Exclusion Criteria:

- Primary care providers who work less than 20% full time equivalent (FTE)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Golberstein, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The original study protocol included a potential second randomization period after six months into the trial. This secondary randomization did not occur, per the recommendation of the Data Monitoring Committee
Units Other Than Participants: primary care clinics
Period: Overall Study
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Started | 126; 10 primary care clinics | 112; 11 primary care clinics | 104; 9 primary care clinics | 131; 11 primary care clinics
Completed | 126; 10 primary care clinics | 112; 11 primary care clinics | 104; 9 primary care clinics | 131; 11 primary care clinics
Not Completed | 0; 0 primary care clinics | 0; 0 primary care clinics | 0; 0 primary care clinics | 0; 0 primary care clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge | Total
Number analyzed (Participants) | 126 | 112 | 104 | 131 | 473
Age, Categorical [Count of Participants; unit: Participants] — Population: Age information was not collected
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 70 | 64 | 66 | 86 | 286
  Male | 49 | 44 | 38 | 42 | 173
  Unkown | 7 | 4 | 0 | 3 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Opioid Prescription Rate
Description: Outcome reported as the percent of Primary Care Appointments (PCAs) at each clinic during which an opioid is prescribed, without currently receiving a non-opioid alternative pain treatment (including a new order for a non-opioid pain treatment).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Number analyzed (Participants) | 123 | 107 | 102 | 127
percent | 0.0159 (0.125) | 0.0141 (0.118) | 0.0161 (0.129) | 0.0120 (0.109)

2. Secondary Outcome: Rate of Non-Opioid Treatment Prescription
Description: Outcome reported as the percent of Primary Care Appointments (PCAs) at each clinic during which a CDC-recommended non-opioid treatment in ordered
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Number analyzed (Participants) | 123 | 107 | 102 | 127
percent | 0.239 (0.426) | 0.227 (0.419) | 0.23 (0.421) | 0.228 (0.419)

3. Secondary Outcome: Opioid Prescription Length
Description: Outcome reported as the mean length of opioid prescription (in days) given during Primary Care Appointments
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Number analyzed (Participants) | 123 | 107 | 102 | 127
Days | 9.63 (18.66) | 11.85 (21.4) | 13.43 (35.86) | 11.75 (25.39)

4. Secondary Outcome: Opioid Prescription MME
Description: Outcome reported as the mean Milligram Morphine Equivalents (MME) of opioid prescriptions given during Primary Care Appointments
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Milligram Morphine Equivalents
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
Number analyzed (Participants) | 123 | 107 | 102 | 127
Milligram Morphine Equivalents | 23.41 (14.9) | 23.89 (18.3) | 21.6 (12.1) | 23.89 (15.9)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | Care as Usual | Choice Architecture Nudge | PMP Integration & Nudge | Choice Architecture Nudge + PMP Integration & Nudge
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04601493/Prot_SAP_000.pdf